CLINICAL TRIAL: NCT03379740
Title: A Single-center, Open-label, Concentration-ranging Study to Investigate the Nicotine Pharmacokinetic Profiles and Pharmacodynamic Effects of the P4M3 Variants
Brief Title: Study to Investigate the Nicotine Pharmacokinetic Profiles and Pharmacodynamic Effects of P4M3 Variants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P4M3-PK-02-US
Record Dates: First submitted 2017-12-01; First posted 2017-12-20 (Actual); Results first posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Vaping; Nicotine Absorption
Keywords: Nicotine-containing product; Alternative to cigarettes
MeSH Terms: conditions — Vaping | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Masking Description: This is an open-label study; however the site (except the pharmacy staff preparing the IPs for administration) will be masked to the randomization sequences until they are assigned. Subjects will not be informed of the complete sequence to which they have been assigned to receive the P4M3 products.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Product Exposure Sequence 1 (Experimental): Subjects will be randomized to follow a sequence of product exposure comprised of :
  Subject's own e-cigarette; P4M3-1.7%; P4M3-1.7%LA; P4M3-3%LA; and P4M3-4%LA
  Interventions: Other: E-cigarette; Other: P4M3-1.7%; Other: P4M3-1.7%LA; Other: P4M3-3%LA; Other: P4M3-4%LA
- Product Exposure Sequence 2 (Experimental): Subjects will be randomized to follow a sequence of product exposure comprised of :
  Subject's own e-cigarette; P4M3-1.7%LA; P4M3-1.7%; P4M3-3%LA; and P4M3-4%LA
  Interventions: Other: E-cigarette; Other: P4M3-1.7%; Other: P4M3-1.7%LA; Other: P4M3-3%LA; Other: P4M3-4%LA

INTERVENTIONS:
Other: E-cigarette — Subject's own e-cigarette
Other: P4M3-1.7% — P4M3 e-liquid concentration of 1.7% nicotine without lactic acid
Other: P4M3-1.7%LA — P4M3 e-liquid concentration of 1.7% nicotine with lactic acid
Other: P4M3-3%LA — P4M3 e-liquid concentration of 3% nicotine with lactic acid
Other: P4M3-4%LA — P4M3 e-liquid concentration of 4% nicotine with lactic acid

SUMMARY:
This is a single-center, open-label, concentration-ranging study to evaluate the nicotine PK profile and PD effects in healthy adult experienced users of closed tank/cartridge e-cigarettes using four different variants of P4M3 (nicotine concentration of 1.7%, 1.7% with 1.1% lactic acid [LA], 3% with 1.1% LA, and 4% with 2% LA) or their own e-cigarettes.

DETAILED DESCRIPTION:
The goal of the study is to evaluate the nicotine concentration profiles and derived PK parameters, subjective effects, behavioral parameters, including puffing topography parameters of P4M3 with four different variants of P4M3, in experienced e-cigarette users after a single-use experience with fixed puffing regime and after ad libitum use of P4M3.

Four variants of P4M3 will be evaluated together with subjects' own e-cigarettes to evaluate the relationship between the e-liquid composition (nicotine concentrations and presence of lactic acid) and the amount of nicotine absorbed, the speed of absorption, and the puffing topography.

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed the informed consent form (ICF) and is able to understand the information provided in the ICF.
* Subject is 21 to 65 years of age, inclusive, at the Screening Visit.
* Subject is a former daily cigarette smoker who smoked at least 100 cigarettes or more in his/her life and ceased smoking at least 3 months prior to the Screening Visit.
* Subject has been using a commercially available, nicotine-containing closed tank/cartridge e-cigarette daily for at least 3 months prior to the Screening Visit.
* Subject has a urine cotinine test ≥200 ng/mL at the Screening Visit and Admission.

Exclusion Criteria:

* Subject has a clinically relevant disease which requires medication which as per the judgment of the Investigator would jeopardize the safety of the subject.
* Subject has abnormal renal function test result or subject with a creatinine clearance <60 mL/minute at the Screening Visit, confirmed on repeat testing.
* Subject has elevated liver function test results at the Screening Visit.
* Subject has bilirubin >1.5X ULN at the Screening Visit.
* Subject has FEV1/FVC <0.7 and FEV1 <80% predicted value at post-bronchodilator spirometry at the Screening Visit.
* Subject has asthma condition at the Screening Visit.
* Subject has received medication within 14 days or within 5 half-lives of the drug (whichever is longer) prior to Admission, which has an impact on cytochrome P450 (CYP) 2A6 activity.
* Subject has a carbon monoxide (CO) breath test ≥ 10 ppm at the Screening Visit or Admission.
* Subject has a body mass index (BMI) <18.5 kg/m2 or BMI ≥35 kg/m2 at the Screening Visit.
* Subject has a positive serology test for human immunodeficiency virus (HIV) 1/2, hepatitis B, or hepatitis C at the Screening Visit.
* Subject has clinically significant ECG findings at the Screening Visit.
* Subject has participated in a clinical study within 3 months prior to the Screening Visit.
* Subject smokes cigarettes or uses other tobacco products.
* Female subject of childbearing potential who is pregnant or breastfeeding.
* Female subject of childbearing potential who does not agree to use an acceptable method of effective contraception..

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Haziza, PhD, Study Chair — Philip Morris Products S.A.; Jonathan Austin, MD, Principal Investigator — High Point Clinical Trials Center
Locations (1):
- High Point Clinical Trials Center, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Product Exposure Sequence 1: Subjects will be randomized to follow a sequence of product exposure comprised of :
  E-cigarette; P4M3-1.7%; P4M3-1.7%LA; P4M3-3%LA; and P4M3-4%LA
  E-cigarette: Subject's own e-cigarette
  P4M3-1.7%: P4M3 e-liquid concentration of 1.7% nicotine without lactic acid
  P4M3-1.7%LA: P4M3 e-liquid concentration of 1.7% nicotine with lactic acid
  P4M3-3%LA: P4M3 e-liquid concentration of 3% nicotine with lactic acid
  P4M3-4%LA: P4M3 e-liquid concentration of 4% nicotine with lactic acid
- Product Exposure Sequence 2: Subjects will be randomized to follow a sequence of product exposure comprised of :
  E-cigarette; P4M3-1.7%LA; P4M3-1.7%; P4M3-3%LA; and P4M3-4%LA
  E-cigarette: Subject's own e-cigarette
  P4M3-1.7%: P4M3 e-liquid concentration of 1.7% nicotine without lactic acid
  P4M3-1.7%LA: P4M3 e-liquid concentration of 1.7% nicotine with lactic acid
  P4M3-3%LA: P4M3 e-liquid concentration of 3% nicotine with lactic acid
  P4M3-4%LA: P4M3 e-liquid concentration of 4% nicotine with lactic acid
Period: Overall Study
Arm/Group | Product Exposure Sequence 1 | Product Exposure Sequence 2
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Product Exposure Sequence 1 | Product Exposure Sequence 2 | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Full Range); unit: years] | 38.3 [22 to 59] | 42.0 [21 to 55] | 40.0 [21 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight (kg) [Mean (Full Range); unit: kg] | 83.95 [65.1 to 120.5] | 70.41 [61.6 to 89.1] | 77.63 [61.6 to 120.5]
Height (cm) [Mean (Full Range); unit: cm] | 178.2 [171 to 186] | 165.0 [149 to 180] | 172.1 [149 to 186]
BMI (kg/m^2) [Mean (Full Range); unit: kg/m^2] | 26.361 [19.40 to 34.94] | 26.174 [21.22 to 34.80] | 26.274 [19.40 to 34.94]

OUTCOME MEASURES:

1. Primary Outcome: Plasma Nicotine Concentration Versus Time Profile
Description: To measure total and background-corrected plasma nicotine concentration versus time profiles from 60 minutes of ad libitum use.
Time Frame: From Day -1 (baseline) to Day 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Subject's Own E-cigarette: Subject's own e-cigarette with e-liquid
- P4M3-1.7%: P4M3 with e-liquid concentrations of 1.7% nicotine without lactic acid
- P4M3-1.7%LA: P4M3 with e-liquid concentrations of 1.7% nicotine with lactic acid
- P4M3-3%LA: P4M3 with e-liquid concentrations of 3% nicotine with lactic acid
- P4M3-4%LA: P4M3 with e-liquid concentrations of 4% nicotine with lactic acid
Arm/Group | Subject's Own E-cigarette | P4M3-1.7% | P4M3-1.7%LA | P4M3-3%LA | P4M3-4%LA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
ng/mL
  10 mins | 4.546 (99.52) | 3.165 (77.27) | 4.167 (119.38) | 7.518 (93.39) | 6.782 (95.57)
  20 mins | 7.235 (103.89) | 5.237 (65.20) | 6.990 (121.67) | 11.92 (65.52) | 9.942 (65.34)
  30 mins | 8.852 (113.80) | 7.808 (62.57) | 8.165 (111.02) | 17.85 (66.05) | 14.65 (60.02)
  40 mins | 10.25 (111.09) | 9.338 (61.00) | 9.852 (99.60) | 20.72 (63.01) | 19.17 (56.21)
  60 mins | 14.46 (80.78) | 13.24 (55.46) | 12.64 (96.63) | 25.53 (62.65) | 25.77 (55.60)
  120 mins | 8.809 (90.18) | 9.356 (69.35) | 7.157 (102.04) | 15.52 (52.34) | 12.76 (50.27)
  240 mins | 4.297 (91.97) | 4.524 (76.68) | 3.311 (91.70) | 7.490 (53.81) | 5.681 (45.33)

2. Primary Outcome: Peak Plasma Nicotine Concentration [cCpeak]
Description: To measure background-corrected peak plasma nicotine concentration [cCpeak] from 60 minutes of ad libitum use.
Time Frame: From Day -1 (baseline) to Day 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Subject's Own E-cigarette | P4M3-1.7% | P4M3-1.7%LA | P4M3-3%LA | P4M3-4%LA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
ng/mL | 14.87 (83.01) | 13.32 (55.65) | 13.05 (98.16) | 26.47 (63.68) | 26.57 (57.34)

3. Primary Outcome: Time to Peak Plasma Nicotine Concentration [Tpeak]
Description: To measure the time to peak plasma nicotine concentration [tpeak] from 60 minutes of ad libitum use.
Time Frame: From Day -1 (baseline) to Day 4
Measure: Median (Full Range); unit: minutes
Arm/Group | Subject's Own E-cigarette | P4M3-1.7% | P4M3-1.7%LA | P4M3-3%LA | P4M3-4%LA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
minutes | 60.000 [30.00 to 65.00] | 60.000 [60.00 to 122.00] | 60.000 [40.00 to 60.00] | 60.000 [30.00 to 60.00] | 60.000 [40.00 to 65.00]

4. Primary Outcome: Background-corrected Trough Plasma Nicotine Concentration [cCtrough]
Description: To measure background-corrected trough plasma nicotine concentration [cCtrough] from 60 minutes of ad libitum use.
Time Frame: From Day -1 (baseline) to Day 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Subject's Own E-cigarette | P4M3-1.7% | P4M3-1.7%LA | P4M3-3%LA | P4M3-4%LA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
ng/mL | 3.492 (98.26) | 2.819 (74.17) | 2.905 (101.32) | 6.032 (73.40) | 4.845 (59.40)

5. Primary Outcome: Background-corrected Average of Plasma Nicotine Concentration [cCaverage]
Description: To measure background-corrected average of plasma nicotine concentration between 0 to 1 hour [cCaverage] from 60 minutes of ad libitum use.
Time Frame: From Day -1 (baseline) to Day 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Subject's Own E-cigarette | P4M3-1.7% | P4M3-1.7%LA | P4M3-3%LA | P4M3-4%LA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
ng/mL | 8.548 (95.38) | 7.302 (55.95) | 7.870 (101.89) | 16.03 (62.01) | 14.48 (55.31)

6. Secondary Outcome: Total and Background-corrected Plasma Nicotine Concentration Versus Time Profiles
Description: To measure the total and background-corrected plasma nicotine concentration versus time profiles of the P4M3 variants and subjects' own e-cigarette from the fixed puffing regimen.
Time Frame: From Day -1 (baseline) to Day 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Subject's Own E-cigarette | P4M3-1.7% | P4M3-1.7%LA | P4M3-3%LA | P4M3-4%LA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
ng/mL
  2 mins | 1.228 (138.63) | 0.7868 (268.65) | 1.620 (117.19) | 2.025 (165.36) | 3.634 (143.44)
  4 mins | 3.158 (107.95) | 1.915 (120.88) | 4.048 (126.28) | 4.817 (113.35) | 7.356 (65.15)
  7 mins | 4.960 (81.41) | 3.992 (77.63) | 5.869 (83.79) | 8.162 (67.20) | 9.905 (69.36)
  10 mins | 4.443 (80.92) | 4.386 (66.40) | 5.232 (72.58) | 7.793 (57.17) | 9.480 (68.97)
  15 mins | 3.810 (71.38) | 3.788 (60.59) | 4.250 (74.72) | 7.251 (57.53) | 8.152 (57.85)
  30 mins | 3.209 (83.26) | 2.704 (98.56) | 3.202 (73.14) | 5.232 (57.79) | 6.203 (66.86)
  60 mins | 2.365 (93.30) | 2.300 (52.26) | 2.352 (71.13) | 3.646 (62.22) | 4.238 (74.41)
  120 mins | 1.579 (96.29) | 1.292 (52.31) | 1.479 (68.44) | 2.074 (65.23) | 2.398 (79.90)
  240 mins | 0.8435 (81.99) | 0.6550 (50.33) | 0.6794 (84.09) | 1.038 (54.59) | 1.183 (74.31)

7. Secondary Outcome: Background-corrected Maximum Plasma Concentration [cCmax]
Description: To measure the background-corrected maximum plasma concentration [cCmax] of the P4M3 variants and subjects' own e-cigarette from the fixed puffing regimen.
Time Frame: From Day -1 (baseline) to Day 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Subject's Own E-cigarette | P4M3-1.7% | P4M3-1.7%LA | P4M3-3%LA | P4M3-4%LA
Number analyzed (Participants) | 15 | 14 | 14 | 15 | 15
ng/mL | 5.402 (78.06) | 5.074 (77.64) | 6.735 (83.39) | 9.437 (63.11) | 11.990 (78.62)

8. Secondary Outcome: Time to the Maximum Concentration [Tmax]
Description: To measure the time to the maximum concentration [tmax] of the P4M3 variants and subjects' own e-cigarette from the fixed puffing regimen.
Time Frame: From Day -1 (baseline) to Day 4
Measure: Mean (Full Range); unit: minutes
Arm/Group | Subject's Own E-cigarette | P4M3-1.7% | P4M3-1.7%LA | P4M3-3%LA | P4M3-4%LA
Number analyzed (Participants) | 15 | 14 | 14 | 15 | 15
minutes | 10.002 [4.00 to 120.00] | 10.002 [4.00 to 60.00] | 7.002 [4.00 to 30.00] | 10.002 [4.00 to 15.00] | 7.002 [2.00 to 15.00]

9. Secondary Outcome: Background-corrected Area Under the Concentration-time Curve [cAUC(0-4h)]
Description: To measure the background-corrected area under the concentration-time curve, which is above the corrected baseline from the start of product use to 4 hours [cAUC(0-4h)], of the P4M3 variants and subjects' own e-cigarette from the fixed puffing regimen.
Time Frame: From Day -1 (baseline) to Day 4
Population: Values below the Lower Limit of Quantification were set to missing.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Subject's Own E-cigarette | P4M3-1.7% | P4M3-1.7%LA | P4M3-3%LA | P4M3-4%LA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
ng*h/mL
  Fixed Regimen: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15
  Fixed Regimen | 7.796 (81.19) | 6.969 (50.19) | 7.679 (66.36) | 11.55 (56.00) | 13.570 (67.10)
  Ad libitum | 33.77 (86.94) | 33.03 (61.44) | 28.64 (96.87) | 60.21 (55.29) | 52.79 (50.19)

10. Secondary Outcome: Subjective Effects of P4M3 Use
Description: Measured with an adapted version of the modified Cigarette Evaluation Questionnaire (adapted mCEQ) within 60 minutes after the ad libitum use session. Assessed on a 7-point scale, ranging from 1 (not at all) to 7 (extremely).
Time Frame: From Day -1 (baseline) to Day 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subject's Own E-cigarette | P4M3-1.7% | P4M3-1.7%LA | P4M3-3%LA | P4M3-4%LA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
score on a scale
  Product Satisfaction | 4.76 (1.058) | 3.62 (1.425) | 3.49 (1.667) | 3.24 (1.165) | 3.04 (1.469)
  Psychological Reward | 3.88 (1.242) | 3.49 (1.396) | 3.13 (1.529) | 3.01 (1.060) | 2.88 (1.207)
  Aversion | 1.77 (0.864) | 1.57 (0.843) | 2.00 (1.036) | 2.37 (1.518) | 2.53 (1.788)
  Enjoyment of Respiratory Tract Sensations | 4.3 (1.23) | 3.2 (1.02) | 3.1 (1.23) | 3.0 (0.93) | 2.9 (1.28)
  Craving Reduction | 4.3 (1.67) | 3.9 (1.25) | 3.7 (1.80) | 3.6 (1.51) | 3.5 (1.85)

11. Secondary Outcome: Area Under the Curve of Craving for an Electronic Cigarette
Description: Measured on a Visual Analogue Scale (VAS) of 0 (no craving) to 100 (strong craving), before and after the fixed puffing regimen and ad libitum use period. (The VAS craving was measured from 0 to 100 on a 100 mm scale.)
  The data below present the Area under the VAS craving score-time curve from the start of product use to 4 hours.
  The area under the curve for VAS craving is an integrated measurement of the VAS craving taking into account several timepoints. AUC was calculated using a trapezoidal rule between timepoints without normalization.
Time Frame: From Day -1 (baseline) to Day 4
Measure: Mean (Standard Deviation); unit: score*hr
Arm/Group | Subject's Own E-cigarette | P4M3-1.7% | P4M3-1.7%LA | P4M3-3%LA | P4M3-4%LA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
score*hr
  Fixed Puffing | 154.8 (120.90) | 134.4 (117.02) | 135.5 (120.61) | 141.8 (105.87) | 124.9 (106.80)
  Ad Libitum | 143.2 (87.05) | 117.9 (84.65) | 119.5 (100.03) | 108.0 (89.93) | 96.9 (90.26)

12. Secondary Outcome: Sensory Parameters (Fixed Puffing Regimen)
Description: Measured with a Sensory Questionnaire (SQ) within 60 minutes after each fixed puffing regimen use period. Response to each question is assessed on a 7-point scale, ranging from 1 (not at all) to 7 (extremely).
Time Frame: From Day 1 to Day 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subject's Own E-cigarette | P4M3-1.7% | P4M3-1.7%LA | P4M3-3%LA | P4M3-4%LA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
score on a scale
  How much did you like the puffs you took? | 4.9 (1.41) | 3.7 (1.34) | 3.7 (1.86) | 3.5 (1.73) | 3.5 (1.25)
  How harsh were the puffs you took? | 3.6 (1.41) | 4.4 (1.30) | 3.2 (1.53) | 4.1 (1.19) | 3.7 (1.54)
  How similar to your own brand were the puffs? | 3.6 (1.81) | 2.3 (1.18) | 2.3 (1.64) | 2.1 (1.07) | 2.3 (1.12)
  Strength of puffs on tongue? | 2.5 (1.13) | 2.8 (1.09) | 2.5 (1.10) | 2.8 (1.21) | 3.0 (1.26)
  Strength of puffs in nose? | 1.9 (0.92) | 2.2 (1.02) | 1.8 (0.81) | 2.2 (0.87) | 2.3 (1.23)
  Strength of puffs in back of mouth & throat? | 3.7 (1.30) | 4.1 (1.19) | 2.9 (1.10) | 3.9 (1.34) | 3.9 (1.51)
  Strength of puffs in windpipe? | 3.3 (1.44) | 4.1 (1.10) | 3.1 (1.08) | 4.1 (1.49) | 3.8 (1.57)
  Strength puffs in chest? | 2.9 (1.13) | 3.5 (1.41) | 2.2 (1.13) | 3.5 (1.83) | 3.2 (1.66)

13. Secondary Outcome: Sensory Parameters (ad Libitum Use)
Description: Measured with a Sensory Questionnaire (SQ) within 60 minutes after each ad libitum use period. Response to each question is assessed on a 7-point scale, ranging from 1 (not at all) to 7 (extremely).
Time Frame: From Day 1 to Day 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subject's Own E-cigarette | P4M3-1.7% | P4M3-1.7%LA | P4M3-3%LA | P4M3-4%LA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
score on a scale
  How much did you like the puffs you took? | 4.7 (1.23) | 3.9 (1.69) | 3.4 (1.64) | 3.6 (1.30) | 3.1 (1.21)
  How harsh were the puffs you took? | 3.1 (1.28) | 3.9 (1.44) | 3.3 (1.45) | 3.3 (1.80) | 3.9 (1.57)
  How similar to your own brand were the puffs? | 3.8 (2.05) | 2.2 (1.09) | 2.1 (1.34) | 2.1 (1.04) | 2.1 (1.00)
  Strength of puffs on tongue? | 3.0 (1.20) | 2.7 (1.05) | 2.5 (1.07) | 2.8 (1.15) | 2.5 (1.17)
  Strength of puffs in nose? | 2.1 (1.04) | 2.0 (0.93) | 2.0 (1.07) | 2.1 (0.89) | 1.8 (0.70)
  Strength of puffs in back of mouth & throat? | 3.5 (0.92) | 3.5 (1.46) | 2.7 (1.17) | 3.4 (1.25) | 3.7 (1.59)
  Strength of puffs in windpipe? | 3.5 (1.00) | 3.9 (1.63) | 2.9 (0.89) | 3.5 (1.31) | 3.7 (1.59)
  Strength puffs in chest? | 3.1 (1.04) | 3.3 (1.55) | 2.9 (1.07) | 3.3 (1.45) | 3.2 (1.58)

14. Secondary Outcome: Human Puffing Topography (HPT) of the P4M3 Variants and the Subjects' Own E-cigarette
Description: Total Puff Volume measured for the P4M3 variants and the subjects' own e-cigarette from the fixed puffing regimen and the 60 minutes ad libitum use.
Time Frame: From Day -1 (baseline) to Day 4
Population: HPT raw data were reviewed for recording errors by personnel independent from the study and accepted or rejected prior to analysis. HPT data with the 'Rejected' status were excluded from the analysis. Consequently, the number of subjects analyzed differ from the overall number of subjects analyzed.
Measure: Geometric Mean (90% Confidence Interval); unit: mL (Total Puff Volume)
Arm/Group | Subject's Own E-cigarette | P4M3-1.7% | P4M3-1.7%LA | P4M3-3%LA | P4M3-4%LA
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
mL (Total Puff Volume)
  Fixed Puffing: number analyzed (Participants) | 13 | 12 | 12 | 13 | 11
  Fixed Puffing | 1103.2913 [896.5624 to 1682.3241] | 1133.2255 [878.6965 to 1844.3455] | 1235.2367 [874.7012 to 2069.0103] | 1139.8381 [857.5359 to 1877.5095] | 935.8970 [739.5238 to 1408.0820]
  Ad Libitum: number analyzed (Participants) | 11 | 13 | 12 | 11 | 10
  Ad Libitum | 2054.8081 [1699.3244 to 2881.0980] | 2752.3456 [2232.0269 to 3976.0701] | 2945.8303 [2516.5662 to 4579.0958] | 2601.0945 [2241.0882 to 3226.3642] | 1934.8479 [1442.3779 to 2951.8173]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the entire study duration of up to 36 days, with individual subject participation of between 15 to 36 days from the signature of the Informed Consent Form (ICF) until the end of the safety follow-up period.
Description: The safety was assessed in the safety population, consisting of all randomized subjects who gave informed consent and had exposure to at least one of the investigational products, including product test, as part of the study.
Groups:
- P4M3-1.7% Product Test: On Admission Day (day -2) all subjects were invited to test the P4M3 product for 10 minutes.
- P4M3-1.7%LA: P4M3 with e-liquid concentrations of 1.7% nicotine with 1.1% lactic acid
- P4M3-3%LA: P4M3 with e-liquid concentrations of 3% nicotine with 1.1% lactic acid
- P4M3-4%LA: P4M3 with e-liquid concentrations of 4% nicotine with 2% lactic acid
Arm/Group | P4M3-1.7% Product Test | Subject's Own E-cigarette | P4M3-1.7% | P4M3-1.7%LA | P4M3-3%LA | P4M3-4%LA
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 1/15 | 2/15 | 0/15 | 4/15 | 2/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P4M3-1.7% Product Test (N=15) | Subject's Own E-cigarette (N=15) | P4M3-1.7% (N=15) | P4M3-1.7%LA (N=15) | P4M3-3%LA (N=15) | P4M3-4%LA (N=15)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrohea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site hypoaesthesia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specify that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belong to the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/40/NCT03379740/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/40/NCT03379740/SAP_001.pdf